CLINICAL TRIAL: NCT03880487
Title: A Randomized, Placebo- and Active-Controlled, Double-Blind, Single and Multiple Ascending Dose Study in Healthy Adults to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of KP-1199
Brief Title: A Single and Multiple Ascending Dose Study in Healthy Subjects to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of KP-1199
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Study was terminated early by sponsor
Sponsor: Kalyra Pharmaceuticals, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: KP-1199-CP-001; CDMRP-OR 160158 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-03-05; First posted 2019-03-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-02

CONDITIONS: Analgesia
Keywords: Phase I, Healthy Adult Participants
MeSH Terms: conditions — Agnosia | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KP-1199 (Experimental)
  Interventions: Drug: KP-1199
- Placebo oral capsules (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- Oxycodone oral capsules (Active Comparator)
  Interventions: Drug: Oxycodone oral capsule

INTERVENTIONS:
Drug: KP-1199 — Single dose and Multiple ascending doses of KP-1199 oral capsules
  Arms: KP-1199
Drug: Placebo oral capsule — Single dose and Multiple dose identical to active treatment but without KP-1199.
  Arms: Placebo oral capsules
Drug: Oxycodone oral capsule — 10 mg Oxycodone Capsules
  Arms: Oxycodone oral capsules

SUMMARY:
This is a Phase I, randomized, placebo and active-controlled, double blind, single and multiple ascending dose study in healthy adults to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of KP-1199

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult 18-45 years of age at time of screening, inclusive.
* Have a body mass index (BMI) between 18.0 and ≤32 kg/m2, inclusive, and a weight of ≥50 kg at screening.
* Be determined to be healthy on the basis of a pre-study physical examination, medical history review, vital sign measurements, and the results of laboratory tests.
* For both male and females: using acceptable method of birth control
* If Female: not-pregnant or not breast feeding and not planning on becoming pregnant
* All prescribed medication must have been stopped at least 14 days prior to admission to the clinical research site. An exception is made for hormonal contraceptives, which may be used throughout the study.
* All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's Wort) must have been stopped at least 14 days prior to admission to the clinical research site.
* Must be adequately informed and understand the nature and risks of the study and must provide written informed consent prior to enrollment at screening.

Exclusion Criteria:

* Subjects who participate in one part of the study are not eligible to participate in subsequent parts of the study.
* Women who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after the follow-up visit.
* Males with female partners who are planning to attempt to become pregnant during this study or within 90 days after the follow-up visit.
* History or evidence of significant clinical or psychiatric disorder, condition, or disease that, in the opinion of the Investigator would pose an unacceptable risk to the subject safety or interfere with the study evaluations, procedures, or completion of the study.
* Documented congenital QT syndrome, and/or corrected QT interval (Fridericia correction; QTcF) at screening or first admission > 450 ms.
* Positive screening test for hepatitis B surface antigen, anti-hepatitis C virus antibodies or anti-human immunodeficiency virus 1 and 2 antibodies.
* History of drug allergy diagnosed by a physician.
* Use of tobacco within 30 days prior to the first study drug administration.
* History of alcohol consumption exceeding 2 standard drinks per day on average.
* Routine or chronic use of more than 0.5 grams of acetaminophen daily.
* History of donation of more than 450 mL of blood within 60 days prior to dosing in the clinical research site or planned donation before 30 days has elapsed since intake of study drug.
* Plasma or platelet donation within 7 days of dosing
* Use of any investigational drug or device within 30 days of the first dose of study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events | Part 1: From Day 1 through Day 6, Part 2: From Day 1 through Day 11, Part 3: From Day 1 through Day 12
  Number of treatment related adverse events as determined by abnormal clinical laboratory tests, vitals signs, physical exam, ECG parameters

SECONDARY OUTCOMES:
Pharmacokinetic Profile of KP-1199 to measure plasma concentration of KP-1199 | Part 1: Day 1 (pre-dose through 4 hours after dose administration), Part 2: (pre-dose through Day 8), Part 3: (pre-dose through Day 7)
  Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetic Profile of KP-1199 to measure Time to Maximum plasma concentration of KP-1199 | Part 1: Day 1 (pre-dose through 4 hours after dose administration), Part 2: (pre-dose through Day 8), Part 3: (pre-dose through Day 7)
  Time to Maximum Plasma Concentration (Tmax)
Pharmacokinetic Profile of KP-1199 to measure area under curve plasma concentration of KP-1199 | Part 1: Day 1 (pre-dose through 4 hours after dose administration), Part 2: (pre-dose through Day 8), Part 3: (pre-dose through Day 7)
  Area Under the Concentration-time Curve Up to Time (t), where t is the last point with concentrations above the lower limit of quantitation (AUC0-t) Area Under the Concentration-time Curve for 1 dosing interval of a multiple dose regimen (AUCtau)
Pharmacokinetic Profile of KP-1199 to measure plasma terminal half-life concentration of KP-1199 | Part 1: Day 1 (pre-dose through 4 hours after dose administration), Part 2: (pre-dose through Day 8), Part 3: (pre-dose through Day 7)
  The Apparent Terminal Elimination Half-life (t1/2)
Pharmacokinetic Profile of KP-1199 to measure the trough plasma concentration of KP-1199 | Part 1: Day 1 (pre-dose through 4 hours after dose administration), Part 2: (pre-dose through Day 8), Part 3: (pre-dose through Day 7)
  Trough Plasma Concentration (Ctrough)
Pharmacodynamic Effects of KP-1199 using Cold Pressor Test to measure pain threshold | Part 3: Day 1, Day 3, Day 5 and Day 7 (pre-dose through 6 hours after dose administration)
  Time to feel first pain ("pain threshold" measured in seconds)
Pharmacodynamic Effects of KP-1199 using Cold Pressor Test to measure pain tolerance | Part 3: Day 1, Day 3, Day 5 and Day 7 (pre-dose through 6 hours after dose administration)
  Time to withdrawal of hand from cold water ("Pain tolerance" in seconds)
Pharmacodynamic Effects of KP-1199 using Cold Pressor Test | Part 3: Day 1, Day 3, Day 5 and Day 7 (pre-dose through 6 hours after dose administration)
  Pain tolerance will be measured at time of hand withdrawal using a 11-point (0-10) Numeric Pain Rating Scale (NPRS) where "0 (no pain) to 10 (worst pain)"
Pharmacodynamic Effects of KP-1199 using Ultraviolet Burn Model (UVB) | Part 3: Day 1, Day 3, Day 5 and Day 7 (pre-dose through 6 hours after dose administration)
  Neurosensory Testing (change in neurosensory assessments of the skin at site of ultraviolet burn)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Bunker, PhD, Study Director — Kalyra Pharmaceuticals, Inc.
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States